CLINICAL TRIAL: NCT02200926
Title: Effects of Slow Loaded and Unloaded Breathing Training
Brief Title: Non-pharmacological Treatment for Essential Isolated Systolic Hypertension in Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Khon Kaen University (Other)
Responsible Party: Principal Investigator, Benjarat Sangthong, Cardiopulmonay research, Faculty of associated medical science, Khon Kaen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BSangthong; change1me (Registry Identifier: Benjarat Sangthong)
Record Dates: First submitted 2014-07-24; First posted 2014-07-25 (Estimated); Last update posted 2016-09-12 (Estimated); Status verified 2016-09

CONDITIONS: Systolic Essential Hypertension

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Experimental): The breathing was performed normally in this groups.
  Interventions: Other: Placebo
- Loaded breathing training (Experimental): subjects will trained to inspire deeply against the resistance setting by using BreathMAX® at the loaded of 18 cmH2O with breathing frequency control at 6 breaths/minute. Breathing pattern will be controlled at duty cycle of 0.4 (inspiratory time = 4 sec and total respiratory time = 10 sec). The training program will be performed at home for 30 minutes/day, 7 days/week for 8 weeks.
  Interventions: Other: Loaded breathing training
- Unloaded breathing training (Experimental): subjects will trained to inspire deeply (no resistance) with breathing frequency control at 6 breaths/minute. Breathing pattern will be controlled at duty cycle of 0.4 (inspiratory time = 4 sec and total respiratory time = 10 sec). The training program will be performed at home for 30 minutes/day, 7 days/week for 8 weeks.
  Interventions: Other: Unloaded breathing training

INTERVENTIONS:
Other: Loaded breathing training — 7 days/weeks, for 8 weeks
  Arms: Loaded breathing training
Other: Unloaded breathing training — 7 days/week, for 8 weeks
  Arms: Unloaded breathing training
Other: Placebo — 7 days/week, for 8 weeks
  Arms: Placebo

SUMMARY:
The previous studies used the slow loaded breathing device for breathing training (Jones et al., 2010). It has been shown that slow loaded breathing training can reduce resting blood pressure and heart rate in essential hypertensive patients. However, this has not been studied in elderly with essential isolated systolic hypertensive patients. Not only highest prevalence of hypertension in Thailand was found in elderly but also physiological changes in the elderly are cause of interest in this special population. It has many advantages to use a slow loaded breathing training in elderly people. Firstly, it is low technology and easily implemented at home. Secondly, it can be practiced almost anytime and anywhere. Thirdly, the orthopedic complications of slow loaded breathing training are minimal. Finally, slow loaded breathing training may be enhancing cardiopulmonary function and other fitness traits, but it out of scope of this study. Moreover, slow loaded breathing exercise by itself should not result in any metabolic adaptation of skeletal muscles, such as the forearm, which had not been trained. If slow loaded breathing training modified some central component of the pressor reflex pathway in a way that single muscle training might work, as suggested above, then loaded breathing training would have a modulating effect on the pressor responses of muscles that had not been trained.

We, therefore, aim to study the effect of slow loaded breathing training by using Breathmax on blood pressure at rest and exercise in elderly with essential isolated systolic hypertension and also investigate the autonomic function and others that may be involved with the changed blood pressure in elderly with essential isolated systolic hypertension. We hypothesized that slow loaded and unloaded breathing training could reduce resting and exercising blood pressure in elderly with essential isolated systolic hypertension.

DETAILED DESCRIPTION:
All subjects will be trained for blood pressure and heart rate measurement at home by using a digital arm blood pressure monitoring for 2 weeks control periods before start breathing training. After 2 weeks, subjects in both breathing training groups will trained to inspire deeply against the resistance setting by using Breathmax at the loaded of 18 centimeter of water (cmH2O) and 0 cmH2O (no resistance) with breathing frequency control at 6 breaths/minute in loaded breathing (LB) and unloaded breathing (ULB) group, respectively. They will rest for 5 seconds after every 6 deep breathing. Breathing pattern will be controlled at duty cycle of 0.4 (inspiratory time = 4 sec and total respiratory time = 10 sec). The paced breathing will be practice using metronome at the laboratory until the subjects can do independently without metronome. The breathing was performed normally in control groups (C). The training program will be performed at home for 30 minutes/day, 7 days/week for 8 weeks.

After 8 weeks of breathing training, the sustainability of breathing training effect will be assessed. Subjects in both breathing training groups (LB and ULB) will be stop breathing training with Breathmax and change to breathing normally. In contrast with the subjects in control group, they will be divided to 2 subgroups. The first subgroup performed loaded breathing training at the loaded of 18 cmH2O. The another subgroup performed unloaded breathing training at the loaded of 0 cmH2O. Breathing frequency will be control at 6 breaths/minute in both subgroups. The training program will be performed at home for 30 minutes/day, 7 days/week for 8 weeks.

Data collection will be carried out for 4 times: (1) before control, (2) before training, (3) after training and (4) after stop training. All measurement will be done in the cardiovascular laboratory room, department of physical therapy, faculty of associated medical sciences. In addition, self measurement of blood pressure and heart rate will be conducted at home every morning after getting up at the same time throughout the study (from week 0 to 18).

ELIGIBILITY:
Inclusion Criteria:

* Essential isolated systolic hypertension (stage I- II, based on recommendations of JNC-VII)
* Good communication

Exclusion Criteria:

* Essential hypertension stage III or secondary hypertension
* History of respiratory disease, heart disease, renal disease, blindness, deafness and cerebrovascular disease.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-07; Primary Completion 2015-11 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Resting blood pressure | 4 months

SECONDARY OUTCOMES:
Heart rate | 4 months
Pulse wave velocity | 4 months
Exercise pressure response | 4 months
Heart rate variability | 4 months
cardiac output | 4 months
Flow-mediated dilatation of brachial artery | 4 months
Forearm limb blood flow | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Benjarat Sangthong, M.Sc., Principal Investigator — Faculty of associated medical science, Khon Kaen University, thailand
Locations (1):
- Faculty of associated medical science, Khon Kaen University, Muang, Changwat Khon Kaen, Thailand

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Jones CU, Sangthong B, Pachirat O. An inspiratory load enhances the antihypertensive effects of home-based training with slow deep breathing: a randomised trial. J Physiother. 2010;56(3):179-86. doi: 10.1016/s1836-9553(10)70023-0. PMID 20795924